CLINICAL TRIAL: NCT02099968
Title: Intensivierte Ernährungs- Und Lebensstilmodifikation Bei Patienten Mit Bluthochdruck Und Kardiometabolischer Risikokonstellation. Eine Zweizentrische Randomisiert-kontrollierte Interventionsstudie über 6 Monate
Brief Title: Comprehensive Lifestyle Modification for Patients With Hypertension and Metabolic Syndrome: a Multicenter Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Kliniken Essen-Mitte (Other); Immanuel Hospital Berlin, Berlin, Germany (Unknown); Charite University, Berlin, Germany (Other); University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Gustav Dobos, Head of Department, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORONA
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive Lifestyle Modification (Experimental)
  Interventions: Behavioral: Comprehensive Lifestyle Modification
- Standard Lifestyle Modification / modified DASH (Active Comparator)
  Interventions: Behavioral: Standard Lifestyle Modification / modified DASH

INTERVENTIONS:
Behavioral: Comprehensive Lifestyle Modification — * Fasting (1st week), followed by:
  * Vegetarian and modified DASH diet (plant-based, low-salt)
  * Aerobic exercise
  * Stress reduction techniques: progressive muscle relaxation, meditation, yoga
  Arms: Comprehensive Lifestyle Modification
Behavioral: Standard Lifestyle Modification / modified DASH — * Modified DASH (vegetarian focused, plant-based, low-salt)
  * Aerobic exercise
  * Stress reduction techniques: progressive muscle relaxation
  Arms: Standard Lifestyle Modification / modified DASH

SUMMARY:
Different forms of diet, e.g. Mediterranean diet, DASH diet, or fasting, have demonstrated efficacy in reducing elevated blood pressure. Moreover, Mediterranean diet, and fasting seem to be effective in improving insulin sensitivity in type 2 diabetes. Further, studies on meditation or mindfulness-based interventions have shown positive effects in patients with hypertension and/or type 2 diabetes. Comprehensive Lifestyle Modification, this is a combination of diet, exercise, and stress management, have improved coronary atherosclerosis. However, no studies have yet investigated the effects of Comprehensive Lifestyle Modification in patients with metabolic syndrome and/or in combination with fasting therapy.

This study is supported by a grant from the Corona-Foundation, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension or antihypertensive medication or subclinical atherosclerosis
* Metabolic syndrome
* Basic mobility

Exclusion Criteria:

* Diabetes type 1
* Insulin bolus therapy
* Coronary artery disease
* Myocardial infarct, pulmonary embolism, or stroke within the past 3 months
* Heart failure
* Peripheral vascular disease
* Chronic kidney disease
* Eating disorder
* Dementia
* Other severe internal disease

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 months
  24-hour ambulatory blood pressure
HOMA Index | 3 months
  Homeostatic Model Assessment

SECONDARY OUTCOMES:
Blood pressure | 3 months, 6 months, 12 months
  24-hour ambulatory blood pressure
Blood pressure | 1 week, 3 months, 6 months, 12 months
  Sphygmomanometer
Pulse wave velocity | 3 months, 6 months, 12 months
  Pulse wave velocity (PWV) is a measure of arterial stiffness
PROCAM | 1 week, 3 months, 6 months, 12 months
  PROCAM risk score
SCORE | 1 week, 3 months, 6 months, 12 months
  SCORE risk score
Waist circumference | 1 week, 3 months, 6 months, 12 months
Weight | 1 week, 3 months, 6 months, 12 months
Blood glucose level | 1 week, 3 months, 6 months, 12 months
Blood insulin level | 1 week, 3 months, 6 months, 12 months
HbA1C | 3 months, 6 months, 12 months
  Longterm parameter for plasma glucose concentration.
Blood creatinine level | 1 week, 3 months, 6 months, 12 months
Total cholesterol | 1 week, 3 months, 6 months, 12 months
LDL cholesterol | 1 week, 3 months, 6 months, 12 months
HDL cholesterol | 1 week, 3 months, 6 months, 12 months
Medication use | 1 week, 3 months, 6 months, 12 months
HADS | 1 week, 3 months, 6 months, 12 months
  Hospital Anxiety and Depression Scale
POMS | 1 week, 3 months, 6 months, 12 months
  Profile of Mood States
CPSS | 3 months, 6 months, 12 months
  Cohen Perceived Stress Scale
SWE | 1 week, 3 months, 6 months, 12 months
  General self-efficacy (Skala zur Allgemeinen Selbstwirksamkeitserwartung)
SF-36 | 3 months, 6 months, 12 months
  Health-related quality of life
MAAS | 3 months, 6 months, 12 months
  Mindfulness Attention Awareness Scale
SCS | 1 week, 3 months, 6 months, 12 months
  Self-Compassion Scale
Lifestyle questionnaire | 3 months, 6 months, 12 months
  Questionnaire on physical activity, stress management, diet
Hair steroid analysis | 6 months, 12 months
  Assessment of long-term glucocorticoid levels in scalp hair.
Bioelectrical impedance analysis | 1 week, 3 months, 6 months, 12 months
  Method for estimating body composition (body fat).
Waist/hip ratio | 1 week, 3 months, 6 months, 12 months
Immunophenotyping | 1 week, 3 months, 6 months
  Assessment of immunological subsets in PBMCs
Intestinal microbiota | 1 week, 3 months, 6 months
  Characterization of gut microbiota.
Metabolomics | 1 week, 3 months
  Assessment of small-molecule metabolite profiles from capillary blood
Gene expression profiling | 1 week, 3 months
  Assessment of gene expression profiles from PBMCs.
Interleukin- 6 | 1 week, 3 months, 6 months, 12 months
CRP | 1 week, 3 months, 6 months, 12 months
Uric acid | 1 week, 3 months, 6 months, 12 months
Insulin-like growth factor (IGF-1) | 1 week, 3 months, 6 months, 12 months
Adverse events | 1 week, 3 months, 6 months, 12 months
  Adverse events
Framingham-Score | 1 week, 3 months, 6 months, 12 months
JBS3-Score | 1 week, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Immanuel Hospital Berlin, Department of Internal and Complementary Medicine, Berlin
  - Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen

REFERENCES:
- [Derived] Maifeld A, Bartolomaeus H, Lober U, Avery EG, Steckhan N, Marko L, Wilck N, Hamad I, Susnjar U, Mahler A, Hohmann C, Chen CY, Cramer H, Dobos G, Lesker TR, Strowig T, Dechend R, Bzdok D, Kleinewietfeld M, Michalsen A, Muller DN, Forslund SK. Fasting alters the gut microbiome reducing blood pressure and body weight in metabolic syndrome patients. Nat Commun. 2021 Mar 30;12(1):1970. doi: 10.1038/s41467-021-22097-0. PMID 33785752